CLINICAL TRIAL: NCT04287465
Title: Comparison of Outcomes in Asleep and Awake DBS With a Directional Electrode
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital District of Helsinki and Uusimaa (Other)
Collaborators: University of Turku (Other)
Responsible Party: Principal Investigator, Maija Koivu, Principal Investigator, Hospital District of Helsinki and Uusimaa
Other Study IDs: HospitalHDU
Record Dates: First submitted 2019-06-25; First posted 2020-02-27 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Parkinson Disease; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To compare the clinical outcome of patients with Parkinson's disease (PD) treated with directional deep brain (dDBS) stimulation undergoing subthalamic deep brain stimulation operation (STN-DBS) under general anesthesia versus local anesthesia.

DETAILED DESCRIPTION:
To compare the clinical outcome of patients with Parkinson's disease (PD) treated with directional deep brain (dDBS) stimulation undergoing subthalamic deep brain stimulation operation (STN-DBS) under general anesthesia versus local anesthesia.

In awake group, 10 patients with Parkinson's disease were treated with St Jude Medical/Abbott Infinity DBS system, and the electrode implantation and testing were performed while the patients were awake. In asleep group, 14 patients with Parkinson's disease were treated with St Jude Medical/Abbott Infinity DBS system, and the electrode implantation were performed while the patients were under general anesthesia. The clinical outcome of the DBS treatment, possible adverse effects and the electrode placement will be compared within these two groups.

ELIGIBILITY:
Inclusion Criteria:

Advanced Parkinson's disease

* The clinical decision of DBS treatment
* The clinical inclusion criteria of DBS treatment:
* drug-resistant tremor
* severe daily motor fluctuations or dyskinesia in despite of the optimal oral medication
* an improvement of UPDRS III scores over 30 % in levodopa challenge test.

Exclusion Criteria:

* The general exclusion criteria for DBS treatment:
* a major depression
* on-going psychosis
* a significant brain atrophy observed in a brain MRI
* a suspicion of atypical parkinsonism
* marked cognitive decline.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with advanced Parkinson's disease and their willingness to undergo DBS operation and treatment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of UPDRS III score | 6 months
  The UPDRS III score (0-60 points) at 6-months' follow-up compared to preoperative UPDRS III score

SECONDARY OUTCOMES:
The change of levodopa equivalent dose, LED | 6 months
  The change of levodopa equivalent dose (LED 0 - 2000 mg) at 6-months' follow-up compared to preoperative LED
Electrode trajectory | 6 months
  The comparison of the actual trajectory of the DBS electrode and the anticipated trajectory of the DBS electrode in both patient groups

CONTACTS AND LOCATIONS:
Overall Officials: Eero Pekkonen, M.D-, Ph.D., Study Director — HUH
Locations (1):
- HUH Meilahti Hospital, department of neurology, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided